CLINICAL TRIAL: NCT06634784
Title: The BONEBRIDGE in Children Below Five Years of Age Premarket Clinical Investigation
Brief Title: Evaluating the Safety of BONEBRIDGE Implants in Children Under Five Years Old: This Study Looks at Children Under Five Who Got BONEBRIDGE BCI 602 Implants. It Collects Information on Any Problems With the Device or the Surgery to See if it is Safe Within the First Year After the Operation.
Acronym: 2023BB006
Status: Active, not recruiting | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023BB006; CIV-24-01-045738 (Other: Bundesinstitut für Arzneimittel und Medizinprodukte)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed; Children Under 5 Years
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural | interventions — Bone Conduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bone Conduction Implant (BCI) — Improvement in hearing using BCI.

SUMMARY:
This study, titled "The BONEBRIDGE in Children Under Five: Premarket Clinical Investigation" (Study ID 2023BB006), looks at kids under five who have received the BONEBRIDGE BCI 602 hearing implant. This observational study, which is both retrospective (looking back) and prospective (looking forward), will take place at multiple hospitals. The main goal is to see if the BONEBRIDGE implant is safe for young children within 12 months after surgery.

Primary Goal: The study's main aim is to collect all information about any bad experiences or issues related to the device and the surgery to check its safety.

Secondary Goals:

Hearing Improvement: Using tests like the Göttinger Speech Intelligibility Test (Word Recognition Scores) to see how much the hearing improves with the implant.

Treatment History: Surgeons will fill out questionnaires about how the treatment went.

Quality of Life: Parents will answer questions about their child's quality of life using the GCBI questionnaire at least 12 months after the implant.

The study will last up to 12 months, including enrolling participants and performing all necessary procedures. The target number of participants includes at least 12 sets of data for safety checks and at least 5 sets of hearing performance data.

By collecting detailed information on any problems and assessing the performance of the BONEBRIDGE implant, this study aims to determine if it is safe and effective for young children.

ELIGIBILITY:
Inclusion Criteria:

Children who received the BONEBRIDGE BCI 602 implant before the age of five and have had the implant for at least 12 months.

Ability to perform the German language test. Willingness and ability to undergo all tests required by the study. Signed and dated informed consent obtained before any study-specific procedure and collection of retrospective data.

Exclusion Criteria:

Inability to perform audiological tests due to psychological, emotional, or related physical disorders.

Failure to meet any inclusion criteria. Any condition that, in the investigator's opinion, poses an increased risk to the patient or prevents full compliance or completion of the study.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 5 years old with BONEBRIDGE BCI 602 implants
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of speech intelligibility using the Göttinger Speech Intelligibility Test. | Day 1
  Hearing Improvement: determined by using the Göttinger Speech Intelligibility Test (Word Recognition Scores). Improvements in hearing with the BONEBRIDGE implant will be evaluated in device aided and unaided condition at least 12 months post-implantation.

SECONDARY OUTCOMES:
Assessment of quality of life using the GCBI questionnaire | Day 1
  Quality of life questionnaires (GCBI) for parents at least 12 months post-implantation.
Evaluation based on treatment history questionnaires for surgeons | Day 1
  Surgeons will complete questionnaires about the treatment history.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Schleswig-Holstein, Klinik für Hals-, Nasen- und Ohrenheilkunde, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No